CLINICAL TRIAL: NCT00945334
Title: Double-blind, Placebo Controlled Trial Comparing Neomycin to Rifaximin Plus Neomycin in the Treatment of Methane Positive Subjects With Constipation-predominant Irritable Bowel Syndrome
Brief Title: Neomycin and Rifaximin Plus Neomycin in Treating Methane Positive Constipation Predominant Irritable Bowel Syndrome
Acronym: C-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark Pimentel, MD (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mark Pimentel, MD, Director, GI Motility Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18709
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome
Keywords: Constipation predominant Irritable Bowel Syndrome
MeSH Terms: interventions — Neomycin; Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Group 1 will receive neomycin (500 mg po bid) and placebo (tid) for 14 days
  Interventions: Drug: Neomycin; Drug: Placebo
- Group 2 (Experimental): Group 2 will receive neomycin (500 mg po bid) and rifaximin (550mg po tid) for 14 days
  Interventions: Drug: Neomycin; Drug: Rifaximin

INTERVENTIONS:
Drug: Neomycin — 500 mg po bid for 14 days
  Other Names: Mycifradin; Neo-Tab; Neo-Fradin
Drug: Placebo — placebo for 14 days tid
  Arms: Group 1
Drug: Rifaximin — 550 mg po tid
  Other Names: Xifaxan
  Arms: Group 2

SUMMARY:
In this study the investigators aim to compare the efficacy of neomycin to a combination of rifaximin and neomycin in the treatment of C-IBS subjects with methane on their breath test. This study will be conducted in collaboration with Dr. John DiBaise at the Mayo Clinic in Scottsdale, AZ and Dr. Satish Rao in Georgia Regents University in Augusta, GA.

ELIGIBILITY:
Inclusion Criteria:

* Rome III positive IBS subjects (18-75 years of age)
* Meet criteria for constipation predominant IBS symptoms including ≤ 3 complete spontaneous bowel movements per week with hard or lumpy stools.
* Presence of detectable methane on single breath sample (≥ 3ppm).
* If subjects are ≥ 50 years old, a colonoscopy had to have been completed within the past 5 years.

Exclusion Criteria:

* Subjects with history of intestinal surgery (except appendectomy or cholecystectomy)
* Recent antibiotic use (within the last 30 days)
* Subjects with known pelvic floor dysfunction
* Pregnancy
* Creatinine level > 1.4
* Poorly controlled/uncontrolled significant medical condition that would interfere with study procedures
* Subjects with hearing loss and/or tinnitus
* History of bowel obstruction
* History of celiac disease
* History of inflammatory bowel disease
* Cirrhosis
* Diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pimentel, MD, FRCP(C), Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Georgia Health Sciences University, Augusta, Georgia

REFERENCES:
- [Background] Pimentel M, Park S, Mirocha J, Kane SV, Kong Y. The effect of a nonabsorbed oral antibiotic (rifaximin) on the symptoms of the irritable bowel syndrome: a randomized trial. Ann Intern Med. 2006 Oct 17;145(8):557-63. doi: 10.7326/0003-4819-145-8-200610170-00004. PMID 17043337
- [Background] Pimentel M, Chatterjee S, Chow EJ, Park S, Kong Y. Neomycin improves constipation-predominant irritable bowel syndrome in a fashion that is dependent on the presence of methane gas: subanalysis of a double-blind randomized controlled study. Dig Dis Sci. 2006 Aug;51(8):1297-301. doi: 10.1007/s10620-006-9104-6. Epub 2006 Jul 11. PMID 16832617

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 19 | 18
Completed | 16 | 15
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (14.3) | 45.5 (16.9) | 42.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Severity of Constipation in Each Arm at Week 1 After Completion of Therapy
Description: Visual analog scale (VAS) score for constipation:
  Severity was rated using a VAS from 0 to 100 units (with 0 = no symptom and 100 = severe symptoms).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 15
units on a scale | 61.2 (24.1) | 28.6 (30.8)

2. Secondary Outcome: Change in Methane From Baseline
Description: Methane output was reported as methane in parts per million (ppm) on breath test:
  Subjects fast for 12 h prior to a breath sample. Breath samples were collected via a Quintron dual bag collecting system and analyzed using a BreathTracker SC. Output was reported as methane in parts per million (ppm) after correction for alveolar sample quality using breath CO2 concentration.
Time Frame: Baseline (Day 0) and Final Visit (Day 44)
Population: Change in breath test methane gas levels: baseline breath test minus final breath test measurement.
Measure: Median (Standard Deviation); unit: parts per million
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 16 | 15
parts per million | 7.5 (9.739557195) | 15 (24.81324182)

ADVERSE EVENTS:
Time Frame: Immediately
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=16) | Group 2 (N=15)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Unwell (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No